CLINICAL TRIAL: NCT07302087
Title: Platelet Serotonin Deficiencies: the Strasbourg Experience
Acronym: SEROTSTG
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9484
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Hemorrhagic Syndrome
Keywords: Hemorrhagic syndrome; Serotonin deficiencies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hemorrhagic syndromes are investigated using algorithms established by reference centers and hemostasis societies.

The investigation of platelet dense granules (nucleotide and serotonin testing) is part of the second-line tests.

It can be performed in cases of platelet aggregation abnormalities in platelet-rich plasma (PRP) suggesting a secretion abnormality, or in cases where the latter is normal, it can be performed if the patient's clinical presentation points to a primary hemostasis abnormality and the clinician wishes to pursue further investigations Intraplatelet serotonin deficiencies are often iatrogenic and may be accompanied by bleeding.

Their impact on platelet function is poorly documented.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥ 18 years old)
* Treated at Strasbourg University Hospital for a hemorrhagic syndrome, suggesting a primary hemostasis abnormality and normal von Willebrand factor, during the period from January 1, 2023, to April 1, 2024.

Exclusion Criteria:

- Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient (≥ 18 years old) treated at Strasbourg University Hospital for a hemorrhagic syndrome, suggesting a primary hemostasis abnormality and normal von Willebrand factor, during the period from January 1, 2023, to April 1, 2024.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Score of ISTH BAT Hemorrhagic Questionnaire | Up to 12 months
  ISTH BAT bleeding questionnaire with its 12-item grid scored from 0 to 4:
  A score ≥ 4 in men or ≥ 6 in women makes the presence of a constitutional hemostasis disorder highly probable

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Ressources et de Compétences des Maladies Hémorragiques Constitutionnelles - CHU de Strasbourg - France, Strasbourg, France